CLINICAL TRIAL: NCT04263181
Title: Identification of AML/MDS Drug Sensitization by in Vivo Chemotherapy Administration
Brief Title: AML/MDS Drug Sensitization by in Vivo Chemotherapy Administration
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Notable Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: 201911201
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cohort 0: -A technical run-in of 5 patients with any of the following:
  * Standard cytarabine/idarubicin induction, includes cytarabine 200 mg/m2 CIVI in 0.9% normal saline over 24 hours for 7 consecutive days (Days 1-7) & idarubicin 12 mg/m2 per day for 3 consecutive days (Days 1-3). Other standard cytarabine-based induction protocols are allowed
  * Decitabine 20 mg/m2/day as a 1-hour infusion on consecutive Days 1-5 or 1-10 of each 28-day cycle.
  * Azacitidine 75 mg/m2/day as a subcutaneous injection on Days 1-7 or on day 1-5 and 8-9 of each 28-day cycle
  * Decitabine 20 mg/m2/day as a 1-hour infusion on consecutive Days 1-5 or 1-10 of each 28-day cycle. Patients will receive venetoclax PO 100 mg on Day 1, 200 mg on Day 2, and 400 mg daily thereafter.
  * Azacitidine 75 mg/m2/day as a 1-hour infusion or by subcutaneous injection on consecutive Days 1-7 or on day 1-5 and 8-9 of each 28-day cycle. Patients will receive venetoclax PO 100 mg on Day 1, 200 mg on Day 2, and 400 mg daily thereafter.
  Interventions: Procedure: Peripheral blood draw; Procedure: Bone marrow aspirate; Procedure: Buccal swab
- Cohort 1: * Patients treated with cytarabine/idarubicin induction therapy
  * Patients will receive a standard cytarabine/idarubicin induction, which includes cytarabine 200 mg/m2 CIVI in 0.9% normal saline over 24 hours for 7 consecutive days (Days 1-7) and idarubicin 12 mg/m2 per day in 0.9% normal saline over 15-30 minutes for 3 consecutive days (Days 1-3). Other standard cytarabine-based induction protocols are allowed (e.g. cytarabine/daunorubicin or Vyxeos).
  Interventions: Procedure: Peripheral blood draw; Procedure: Bone marrow aspirate; Procedure: Buccal swab
- Cohort 2: * Patients treated with decitabine
  * Patients will receive decitabine 20 mg/m2/day as a 1-hour infusion on consecutive Days 1-5 or 1-10 (per treating physician discretion) of each 28-day cycle.
  Interventions: Procedure: Peripheral blood draw; Procedure: Bone marrow aspirate; Procedure: Buccal swab
- Cohort 3: * Patients treated with azacitidine
  * Patients will receive azacitidine 75 mg/m2/day as a subcutaneous injection on Days 1-7 or on day 1-5 and 8-9 (per treating physician discretion) of each 28-day cycle
  Interventions: Procedure: Peripheral blood draw; Procedure: Bone marrow aspirate; Procedure: Buccal swab
- Cohort 4: * Patients treated with decitabine + venetoclax
  * Patients will receive decitabine 20 mg/m2/day as a 1-hour infusion on consecutive Days 1-5 or 1-10 (per treating physician discretion) of each 28-day cycle. Patients will receive venetoclax PO 100 mg on Day 1, 200 mg on Day 2, and 400 mg daily thereafter.
  Interventions: Procedure: Peripheral blood draw; Procedure: Bone marrow aspirate; Procedure: Buccal swab
- Cohort 5: * Patients treated with azacitidine + venetoclax
  * Patients will receive azacitidine 75 mg/m2/day as a 1-hour infusion or by subcutaneous injection on consecutive Days 1-7 or on day 1-5 and 8-9 (per treating physician discretion) of each 28-day cycle. Patients will receive venetoclax PO 100 mg on Day 1, 200 mg on Day 2, and 400 mg daily thereafter.

INTERVENTIONS:
Procedure: Peripheral blood draw — * All cohorts will have peripheral blood drawn at baseline no more than 4 days prior to the first dose of chemotherapy and must also occur before the first dose of chemotherapy
  * Cohort 0 or 1 - peripheral blood draw on Day 2
  * Cohorts 0, 2, 3, 4 and 5 - peripheral blood draw on Day 3
  * Cohort 0 or 1 - peripheral blood draw on Day 35 (at count recovery)
  * Cohorts 0, 2, 3, 4, and 5 - peripheral blood draw on Cycles 2 or 3 and 4 or 5, Day 28
  Groups: Cohort 0; Cohort 1; Cohort 2; Cohort 3; Cohort 4
Procedure: Bone marrow aspirate — * Cohort 0 or 1 - bone marrow aspirate on Day 14
  * Cohort 0 or 1 - bone marrow aspirate on Day 35 (at count recovery)
  * Cohorts 0, 2, 3, 4, and 5 - bone marrow aspirate on Cycles 2 or 3 and 4 or 5, Day 28
  Groups: Cohort 0; Cohort 1; Cohort 2; Cohort 3; Cohort 4
Procedure: Buccal swab — * Cohort 0 or 1 - buccal swab on Day 35 (at count recovery)
  * Cohorts 0, 2, 3, 4, and 5 - buccal swab on Cycle 2 or 3 and 4 or 5, Day 28
  Groups: Cohort 0; Cohort 1; Cohort 2; Cohort 3; Cohort 4

SUMMARY:
In this study, the investigators will explore the feasibility of ex vivo drug screening to predict sensitivity to chemotherapy resistance and to identify novel synergy between chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS)
* Peripheral blood blasts > 1%
* Peripheral white blood cell count > 1,000/µl.
* Age ≥ 18 years
* Anticipated treatment with any of the following regimens (Cohort 0) or:

  * Cohort 1: A standard induction protocol with infusional cytarabine
  * Cohort 2: Decitabine (either 5-day or 10-day regimens)
  * Cohort 3: Azacitidine (either intravenous or subcutaneous administration)
  * Cohort 4: Decitabine (either 5-day or 10-day) + venetoclax
  * Cohort 5: Azacitidine (either intravenous or subcutaneous administration on 7 day or 5+2+2 schedule) + venetoclax
* Patients may receive these therapies as part of other on-going clinical trials or as standard of care treatment.
* Patients in Cohort 1 may receive SOC midostaurin or gemtuzumab ozogamicin, provided these start after the Day 2 sample is collected. Patients in Cohort 1 may receive a standard combination of cytarabine/idarubicin, cytarabine/daunorubicin, or Vyxeos, a liposomal formulation of cytarabine and daunorubicin.
* ECOG performance status ≤ 3
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Pregnant or currently nursing
* Prior chemotherapy with hypomethylating agents
* Known history of positive HIV serology.
* Known positive Hepatitis C serology.
* Patient must not have received any chemotherapy within 7 days of enrollment, and any acute treatment-related toxicities must have returned to baseline. Patients may have received hydrea as long as they fulfill peripheral blood blast and peripheral WBC inclusion criteria. Prior TKI therapy is allowed, but must be discontinued within 3 days of baseline blood collection.
* Currently receiving any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -The study population consists of patients seen at Siteman Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Determine whether ex vivo drug sensitivity obtained for Day 0 ex vivo treatments for all cohorts as measured by a 384 well high throughput flow-based viability assay correlates with clinical assay | 90 days

SECONDARY OUTCOMES:
Ex vivo drug sensitivity obtained for Day 0 ex vivo treatments as measured by a 384 well high throughput flow-based viability assay correlates with molecular responses as measured by founding clone mutation reduction <2% and exome sequencing | 90 days
Determine whether an increase in ex vivo drug resistance on day 2 (cohorts 0 or 1) or day 3 (cohorts 2, 3, 4 and 5), as measured by a 384 well high-throughput flow-based viability assay, correlates with reduced clinical responses | 90 days
Determine whether reduced ex vivo drug sensitivity on day 2 (cohorts 0 or 1) or day 3 (cohorts 2, 3, 4, and 5), as measured by a 384 well high throughput flow-based viability assay, correlates with reduced molecular responses | 90 days
Determine whether reduced drug ex vivo drug sensitivity on day 2 (cohorts 0 or 1) or 3 (cohorts 2, 3, 4, and 5), as measured by a 384 well high throughput flow-based viability assay, correlates with reduced disease-free survival | 1 year
Determine whether reduced ex vivo drug sensitivity, as measured by a 384 well high throughput flow-based viability assay, correlates with reduced survival | 1 year
Determine whether in vivo chemotherapy leads to increased ex vivo sensitivity to any class of drugs in more than 20% of patients treated on any study arm as measured by a 384 well high throughput flow-based viability assay | Day 3
Determine whether decitabine and azacitidine are associated with overlapping or unique profiles in drug sensitivity changes as measured by a 384 well high throughput flow-based viability assay | Day 3
Determine whether ex vivo drug sensitivity, as measured by a 384 well high throughput flow-based viability assay, correlates with the presence of clinically available mutations, as measured by exome sequencing | 90 days
Determine whether MDS and AML have overlapping or unique profiles in ex vivo drug sensitivity, as measured by a 384 well high throughput flow-based viability assay | Day 0
Determine whether MDS and AML have overlapping or unique profiles in ex vivo drug sensitivity as measured by a 384 well high throughput flow-based viability assay | Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Meagan Jacoby, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Blood, buccal cells, and data will be shared. The researchers may be doing research at Washington University, at other research centers and institutions, or industry sponsors of research. Data may also be shared with large data repositories. The researchers may be doing research in areas similar to this research or in other unrelated areas.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years following article publication.
Access Criteria: Proposals should be submitted directly to jwelch@wustl.edu.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu